CLINICAL TRIAL: NCT03911817
Title: Impact of Midodrine Administration on the Clinical Outcome of Septic Shock Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina hussein ahmed eladly, clinical pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 169
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Septic Shock
Keywords: Midodrine; Septic shock; Norepinephrine; Weaning
MeSH Terms: conditions — Shock, Septic | interventions — Midodrine

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV vasopressor (No Intervention): Will receive IV vasopressor infusion only
- Midodrine (Active Comparator): Will receive midodrine in addition to IV vasopressor infusion
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — The oral vasoactive drug (Midodrine) at a dose of 10-20 mg every 8 hours will be used in one arm .After the blood pressure goal is met for more than 24 hours without IV vasopressor ,midodrine will be discontinued prior to discharge
  Arms: Midodrine

SUMMARY:
1. Assess the impact of midodrine administration on weaning of IV vasopressors
2. Assess the cost effectiveness of using midodrine in critically ill patients

DETAILED DESCRIPTION:
A prospective randomized controlled clinical trial on total 60 critically ill patients admitted to critical care medicine department with indication to IV vasopressor due to septic shock on admission or during intensive care unit stay and they are randomly assigned to either of 2 groups as follows

1. Group 1(n=30):will receive IV vasopressor infusion only
2. Group 2(n=30):will receive midodrine in addition to IV vasopressor infusion

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-80)years
2. Hypotensive (systolic blood pressure<90mm Hg)and require IV vasopressor for more than 24 hours
3. Require IV vasopressor at rate < 8mcg/min and unable to wean for >24 hours

Exclusion Criteria:

1. Severe organic heart disease (ejection fraction <30 percent due to higher risk of arrythmia)
2. Bradycardia (HR<50 b/m)due to higher likelihood of symptomatic bradycardia
3. Chronic kidney disease (serum creatinine >2mg/dl) as midodrine and its active metabolites are almost completely execreated in urine
4. Thyrotoxicosis
5. Known allergy to midodrine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Time of weaning of IV vasopressor in both groups | Starting from date of randomization till stop of IV vasopressor completely or date of death from any cause,whichever came first,assessed up to 30 days
  measure duration needed to completely stop IV vasopressor in both groups and the impact of adding midodrine on that duration

SECONDARY OUTCOMES:
ICU length of stay | Starting from date of randomization until ICU discharge or date of death from any cause,whichever came first,assessed up to 30 days
  total duration of patient stay in ICU
Time to ICU discharge after IV vasopressor discontinuation | Starting from discontinuation of IV vasopressor until time to ICU discharge or date of death from any cause ,whichever came first,assessed up to 30 days
  measure duration from IV vasopressor stop till ICU discharge or death
Time to ICU discharge after midodrine initiation | Starting from midodrine initiation until ICU discharge or date of death from any cause,whichever came first,assessed up to 30 days
  measure duration from midodrine start till ICU discharge or death
Mortality | Up to 30 days
  measure if patient die or discharge from the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa ELwakeel, PhD, Principal Investigator — Ain Shams University
Locations (1):
- Critical Care Medicine Department - Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Anstey MH, Wibrow B, Thevathasan T, Roberts B, Chhangani K, Ng PY, Levine A, DiBiasio A, Sarge T, Eikermann M. Midodrine as adjunctive support for treatment of refractory hypotension in the intensive care unit: a multicenter, randomized, placebo controlled trial (the MIDAS trial). BMC Anesthesiol. 2017 Mar 21;17(1):47. doi: 10.1186/s12871-017-0339-x. PMID 28327122
- [Background] Whitson MR, Mo E, Nabi T, Healy L, Koenig S, Narasimhan M, Mayo PH. Feasibility, Utility, and Safety of Midodrine During Recovery Phase From Septic Shock. Chest. 2016 Jun;149(6):1380-3. doi: 10.1016/j.chest.2016.02.657. Epub 2016 Mar 4. PMID 26953217